CLINICAL TRIAL: NCT01546909
Title: Antibody Persistence in 11 to 13-year-old Children Previously Vaccinated at 6 Years Old With Either REVAXIS or DT Polio, and Immune Response to a Booster Dose of TETRAVAC-ACELLULAIRE
Brief Title: Antibody Persistence to REVAXIS or DT Polio and Immune Response to TETRAVAC-ACELLULAIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RVX01C
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diphtheria; Tetanus; Poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TETRAVAC-ACELLULAIRE (Experimental)
  Interventions: Biological: Diphtheria, tetanus, polio and pertussis vaccination

INTERVENTIONS:
Biological: Diphtheria, tetanus, polio and pertussis vaccination — 1 dose of TETRAVAC-ACELLULAIRE (0.5 mL) at Day 0

SUMMARY:
PRIMARY OBJECTIVES

* To describe in 11 to 13-year-old children previously vaccinated with either REVAXIS or DT Polio at 6 years of age the antibody persistence against diphtheria, tetanus, and poliovirus types 1, 2 and 3
* To describe one month after a booster dose of TETRAVAC-ACELLULAIRE the immune responses against diphtheria, tetanus, and poliovirus types 1, 2 and 3

SECONDARY OBJECTIVES

* To describe other parameters of the antibody persistence against diphtheria, tetanus and poliomyelitis antigens
* To describe other parameters of the immune responses to diphtheria, tetanus and poliomyelitis antigens one month after a booster dose of TETRAVAC-ACELLULAIRE
* To describe the safety profile of a booster dose of TETRAVAC-ACELLULAIRE

ELIGIBILITY:
Inclusion Criteria:

* Healthy child 11 to 13 years of age previously vaccinated in Study F05-TdI-301

Exclusion Criteria:

* Immunization against diphtheria, tetanus, pertussis and/or poliomyelitis beyond Study F05-TdI-301
* Previous clinical or bacteriological diagnosis of diphtheria, tetanus, pertussis or poliomyelitis
* Known or suspected immune dysfunction
* Receipt of medications / vaccination that may interfere with study assessments
* Known true hypersensitivity to any of the vaccine components or to a vaccine containing the same substances
* Known personal history of encephalopathy, seizure disorder or progressive, evolving or unstable neurological condition
* Thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection
* Any medical condition that might interfere with the evaluation of the study objectives
* Febrile illness

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an anti-diphtheria concentration ≥0.01 IU/mL | Pre-booster dose (Day 0)
Proportion of subjects with an anti-tetanus concentration ≥0.01 IU/mL | Pre-booster dose (Day 0)
Proportion of subjects with an anti-polio type 1 titer ≥ 8 (1/dilution) | Pre-booster dose (Day 0)
Proportion of subjects with an anti-polio type 2 titer ≥ 8 (1/dilution) | Pre-booster dose (Day 0)
Proportion of subjects with an anti-polio type 3 titer ≥ 8 (1/dilution) | Pre-booster dose (Day 0)
Proportion of subjects with an anti-diphtheria concentration ≥0.1 IU/mL | 1 month post-booster dose
Proportion of subjects with an anti-tetanus concentration ≥0.1 IU/mL | 1 month post-booster dose
Proportion of subjects with an anti-polio type 1 titer ≥8 (1/dilution) | 1 month post-booster dose
Proportion of subjects with an anti-polio type 2 titer ≥8 (1/dilution) | 1 month post-booster dose
Proportion of subjects with an anti-polio type 3 titer ≥8 (1/dilution) | 1 month post-booster dose

SECONDARY OUTCOMES:
Geometric mean titer for diphtheria | Pre-booster (Day 0) and 1 month post-booster dose
Geometric mean titer for tetanus | Pre-booster (Day 0) and 1 month post-booster dose
Geometric mean titer for polio type 1 | Pre-booster (Day 0) and 1 month post-booster dose
Geometric mean titer for polio type 2 | Pre-booster (Day 0) and 1 month post-booster dose
Geometric mean titer for polio type 3 | Pre-booster (Day 0) and 1 month post-booster dose
Solicited injection site and solicited systemic reactions | From Day 0 to Day 7 post vaccination
Unsolicited injection site reactions and unsolicited systemic adverse events | From Day 0 to Day 28 days post vaccination
Serious adverse events | From signature of informed consent up to last study visit of the subject

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (45):
- France (45):
  - SPMSD Investigational Site 120, Angers
  - SPMSD Investigational Site 103, Arras
  - SPMSD Investigational Site 155, Asnières
  - SPMSD Investigational Site 125, Bersée
  - SPMSD Investigational Site 121, Besançon
  - SPMSD Investigational Site 141, Besançon
  - SPMSD Investigational Site 124, Blois
  - SPMSD Investigational Site 161, Blois
  - SPMSD Investigational Site 194, Boulogne-Billancourt
  - SPMSD Investigational Site 148, Brest
  - SPMSD Investigational Site 117, Caen
  - SPMSD Investigational Site 147, Caen
  - SPMSD Investigational Site 163, Champdeniers
  - SPMSD Investigational Site 135, Châlons-en-Champagne
  - SPMSD Investigational Site 145, Chigny-les-Roses
  - SPMSD Investigational Site 157, Cholet
  - SPMSD Investigational Site 101, Clamart
  - SPMSD Investigational Site 160, Collombey Les Belles
  - SPMSD Investigational Site 162, Collombey Les Belles
  - SPMSD Investigational Site 139, Dax
  - SPMSD Investigational Site 193, Draguignan
  - SPMSD Investigational Site 106, Essey-lès-Nancy
  - SPMSD Investigational Site 123, Essey-lès-Nancy
  - SPMSD Investigational Site 164, Essey-lès-Nancy
  - SPMSD Investigational Site 136, Floirac
  - SPMSD Investigational Site 114, Frouard
  - SPMSD Investigational Site 150, Haguenau
  - SPMSD Investigational Site 113, Illkirch-Graffenstaden
  - SPMSD Investigational Site 197, Le Havre
  - SPMSD Investigational Site 198, Le Havre
  - SPMSD Investigational Site 107, Lingolsheim
  - SPMSD Investigational Site 115, Louverné
  - SPMSD Investigational Site 140, Manduel
  - SPMSD Investigational Site 116, Maromme
  - SPMSD Investigational Site 153, Marseille
  - SPMSD Investigational Site 134, Montpellier
  - SPMSD Investigational Site 129, Nogent-sur-Marne
  - SPMSD Investigational Site 133, Ostwald
  - SPMSD Investigational Site 128, Poitiers
  - SPMSD Investigational Site 130, Pont-à-Mousson
  - SPMSD Investigational Site 151, Quimper
  - SPMSD Investigational Site 102, Rouen
  - SPMSD Investigational Site 110, Rouen
  - SPMSD Investigational Site 199, Rouen
  - SPMSD Investigational Site 152, Saint-Ouen